CLINICAL TRIAL: NCT07069959
Title: Early Assessment of Quadriceps Muscle Recovery by Dynamometry and 3D Ultrasound in Intensive Care Patients Under Invasive Mechanical Ventilation: A Monocentric and Prospective Study.
Brief Title: Early Assessment of Quadriceps Muscle Recovery by Dynamometry and 3D Ultrasound in Intensive Care Patients Under Invasive Mechanical Ventilation
Acronym: DYNAMOREA
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0138
Record Dates: First submitted 2025-06-24; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Intensive Care Unit Acquired Weakness; Muscle Weakness
Keywords: dynamometry; muscle weakness; intensive care; functional recovery; invasive mechanical ventilation; 3D ultrasound
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients under invasive mechanical ventilation in the ICU: This group includes patients admitted to the Intensive Care Unit (ICU) at the CHU of Nantes, treated with invasive mechanical ventilation. The study aims to evaluate the early recovery of quadriceps muscle strength in these patients, using non-invasive, pain-free assessment methods. The cohort will consist of approximately 100 patients over one year, with data collected via the medical record and strength measurements performed by physical therapists.
  Interventions: Other: Early assessment of quadriceps muscle strength

INTERVENTIONS:
Other: Early assessment of quadriceps muscle strength — Patients will undergo non-invasive assessment of quadriceps muscle strength using manual dynamometry and 3D ultrasound. These assessments will be conducted regularly during their ICU stay to evaluate early recovery. The intervention is part of routine patient care and does not involve additional treatments or procedures.

SUMMARY:
Patients in intensive care often develop acquired muscle weakness (ICUAW or Intensive Care Unit Acquired Weakness) due to immobilization and muscle atrophy. Early mobilization can help reduce weakness and improve functional recovery, but practices vary. Muscle strength assessment, particularly using the MRC (Medical Research Council) score, is crucial, though it has precision limitations. Additional methods, such as manual dynamometry and functional scales, are needed to better track muscle recovery. The quadriceps, important for function, requires early evaluation, but there is a lack of specific data in intensive care to predict medium-term functional recovery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 18 years
* Hospitalized in an ICU
* Treated with invasive mechanical ventilation (MV) for at least 4 days during their stay (may be extubated at the time of inclusion)
* Conscious and cooperative patients: ability to respond appropriately to the following commands: open and close eyes, look at me, nod your head, stick out your tongue, raise your eyebrows when I count to five
* MRC score ≥ 3/5 for the "Leg Extension" function on either the left or right side
* Informed consent obtained (no opposition)

Exclusion Criteria:

* Pregnant or breastfeeding women
* Fracture or amputation of a lower limb
* Acute or chronic brain or spinal cord injury responsible for hemiplegia or paraplegia
* Unstable spinal injury
* Neurodegenerative or chronic neurological disease
* Guillain-Barré Syndrome
* Myasthenia Gravis
* Acute deep vein thrombosis of the lower limbs treated within the last 48 hours
* Pre-existing motor deficit in a lower limb before the ICU stay, of any cause
* Incarcerated or legally protected individuals (guardianship, curatorship)
* Individuals without social protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adults (aged >18 years) admitted to the ICU and treated with invasive mechanical ventilation for at least 4 days. Participants must be conscious, cooperative, and have an MRC score ≥ 3/5 for "Leg Extension" on either side. Informed consent or no objection is required. Exclusion criteria include pregnancy, neurological disorders, lower limb injuries, or conditions preventing safe participation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Describe the evolution of quadriceps muscle recovery using manual dynamometry in patients under invasive mechanical ventilation in the ICU. | 3 months
  This study aims to describe the evolution of quadriceps muscle recovery in ICU patients under invasive mechanical ventilation, using manual dynamometry as a measurement tool. The recovery will be assessed periodically throughout the ICU stay to evaluate early muscle strength recovery.
Description of the evolution of the recovery of the rectus femoris muscle using 3D ultrasound in ICU patients treated with invasive mechanical ventilation. | 3 months after ICU discharge
  Change in the volume of the rectus femoris muscle measured by 3D ultrasound.

SECONDARY OUTCOMES:
Estimate the average value of the FMQ | From inclusion to 3 months post-ICU discharge
  Measure the FMQ (Quadriceps Muscle Strength ) at multiple key time points to estimate recovery and muscle strength progression.
To study the correlation between FMQ values and other muscular and functional scores on the same day. | From inclusion to 3 months post-ICU discharge
  Correlate FMQ with other muscular and functional scores
Study the differences in muscle strength between right and left FMQ values on the same day | From inclusion to 3 months post-ICU discharge
  Compare right and left side FMQ measurements to assess potential asymmetries.
Study the correlation between FMQ at inclusion and the time until extubation, when the patient was still intubated at inclusion | From inclusion to the day of extubation, an average of 7 days
  Investigate if FMQ at inclusion can predict extubation time in intubated patients.
Study the correlation between FMQ at inclusion and the ability to achieve verticalization for patients who could stand before ICU discharge | From inclusion to ICU discharge, an average of 10 days
  Examine if FMQ at inclusion is predictive of the ability to achieve verticalization during the ICU stay.
Study the correlation between FMQ at inclusion and the ability to take the first steps for patients who were able to walk before ICU discharge | From inclusion to ICU discharge, an average of 10 days
  Assess whether FMQ at inclusion predicts the ability to take first steps during the ICU stay.
Search for an association (survival model) between FMQ (Nm/kg) measured on the day of inclusion and the time (in days) between inclusion and the first steps taken successfully. | 3 months post-ICU discharge
  Study the presence of a link between FMQ (obtained on the day when the patient discharge criteria) and VFMQ (obtained between the day of inclusion and the day the patient inclusion and the day on which the patient meets the criteria for discharge from intensive care) and the patient's functional capacity at the 3-month post-resuscitation consultation. post-resuscitation, linked to an assessment of physical activity during this period. carried out during this period.
Examine how FMQ and VFMQ correlate with strength and functional measures at follow-up, and how physical activity impacts recovery. | 3 months post-ICU discharge
  To study the presence of a link between FMQ (obtained on the day the patient meets the criteria for discharge from intensive care) / VFMQ (obtained between the day of inclusion and the day the patient meets the criteria for discharge from intensive care) and the strength measurement scores obtained during the consultation 3 months after discharge from intensive care, linked to an assessment of physical activity carried out during this period. during this period.
Description of the recovery of the anterior tibial muscle using 3D ultrasound in ICU patients treated with invasive mechanical ventilation. | 3 months after ICU discharge
  Change in the volume of the anterior tibial muscle measured by 3D ultrasound.
Correlation between changes in rectus femoris volume and functional recovery. | 3 months after ICU discharge
  Correlation between volume changes in rectus femoris muscle and functional recovery (between ICU discharge and 3 months post-ICU discharge).
Correlation between changes in anterior tibial muscle volume and functional recovery. | 3 months after ICU discharge
  Correlation between volume changes in the anterior tibial muscle and functional recovery (between ICU discharge and 3 months post-ICU discharge).
Correlation between changes in rectus femoris volume and muscle strength assessment tools. | 3 months after ICU discharge
Correlation between changes in anterior tibial muscle volume and muscle strength assessment tools. | 3 months after ICU discharge
  Correlation between volume changes in the anterior tibial muscle and muscle strength.
Link between rectus femoris volume and functional recovery. | at ICU discharge, an average of 10 days
  Link between rectus femoris volume and functional recovery (at ICU discharge)
Link between rectus femoris volume and functional recovery. | 3 months after ICU discharge
  Link between rectus femoris volume and functional recovery (at 3 months post-ICU discharge)
Link between anterior tibial muscle volume and functional recovery. | at ICU discharge, an average of 10 days
  Link between anterior tibial muscle volume and functional recovery (at ICU discharge)
Link between anterior tibial muscle volume and functional recovery. | 3 months after ICU discharge
  Link between anterior tibial muscle volume and functional recovery (at ICU discharge)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: Undecided